CLINICAL TRIAL: NCT04016857
Title: Effects of Remote Ischemic Preconditioning on Renal Outcomes Following Lower Limb Revascularization
Brief Title: Remote Ischemic Preconditioning During Lower Limb Revascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Alberto Noto, Professor of Anaesthesia, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UMEANE1
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Preconditioning; Acute Kidney Injury; Limb Ischemia
Keywords: remote ischemic preconditioning; lower limb revascularization; TIMP-2; IGFBP-7
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: patients were randomly assigned in 1:1 ratio to either control group or RIPC using computerized randomization table
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The RIPC procedure were performed in the ward before going to operating room, and this is blinded to Investigators and surgical case anesthesiologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC Group (Experimental): Remote ischemic preconditioning
  Interventions: Procedure: RIPC
- Control Group (Sham Comparator): Sham remote ischemic preconditioning
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: RIPC — 4 cycles of 5-min inflation to 200 mmHg followed by 5-min deflation of arm cuff
  Arms: RIPC Group
Procedure: Control — deflated cuff placed on the left arm for 40 min
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the role of remote ischemic preconditioning (RIPC) in preventing acute kidney injury after lower limb revascularization.

Remote ischemic preconditioning(RIPC) is a simple, cost-free and non invasive procedure (transient upper limb ischemia/reperfusion) that could provide organ protection (Heart, Brain and Kidney) following ischemia injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for open limb revascularization

Exclusion Criteria:

* Peripheral vascular disease affecting upper limbs
* Chronic kidney disease in stage 4 or 5 (eGFR<30 ml/min/1,73m2)
* Patients underwent contrast-enhanced radiological exams in the previous 7 days
* Treatment with glibencamide or prostaglandins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
AKI | 72 Hours
  the incidence of Acute Kidney Injury, defined as absolute rise of ≥ 0.3 mg/dL and/or a relative increase of 25% in serum creatinine compared to preoperative
AKI | 72 Hours
  the incidence of Acute Kidney Injury, defined as decrease of 35% in GFR compared to preoperative.

SECONDARY OUTCOMES:
AKI Risk Score | 24 Hours
  the incidence of Acute Kidney Injury, defined as increase od 0.3 in Aki risk score (TIMP-2 * IGFBP-7)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Noto, MD, PhD, Principal Investigator — University of Messina
Locations (1):
- A.O.U. G.Martino - University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: No